CLINICAL TRIAL: NCT03055390
Title: Study the Effect of Intravenous Hyoscine Butylbromide Injection on the Duration and Progress of First Stage Labour in High Risk Women
Brief Title: Effect of Intravenous Hyoscine Butylbromide Injection on Labour in High Risk Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 158
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Vaginal Delivery
Keywords: hyoscine butylbromide; progress of labor; duration of labor
MeSH Terms: interventions — Butylscopolammonium Bromide; 2,3-dioleyloxy-N-(2-(sperminecarboxamido)ethyl)-N,N-dimethyl-1-propanaminium trifluoroacetate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Placebo Comparator): They received two ml of normal saline intravenously as a placebo
  Interventions: Drug: placebo
- 20 mg hyoscine butylbromide (Active Comparator): They received (20mg) hyoscine butylbromide (one ml HBB+ one ml saline) intravenously
  Interventions: Drug: hyoscine butylbromide
- 40 mg hyoscine butylbromide (Active Comparator): They received (40mg) hyoscine butylbromide (one ml HBB+ one ml saline) intravenously
  Interventions: Drug: hyoscine butylbromide

INTERVENTIONS:
Drug: hyoscine butylbromide — Intravenous administration of hyoscine butylbromide during first stage of labor
  Other Names: Dospa
  Arms: 20 mg hyoscine butylbromide; 40 mg hyoscine butylbromide
Drug: placebo — 2ml of saline intravenous
  Other Names: saline
  Arms: Control

SUMMARY:
A case control trial Patients who meet the inclusion criteria were asked to participate in the study and a written consent was obtained from each patient after explaining thoroughly the nature and the scope of the study.

Patients were divided into three equal groups:

Group A: included 40 pregnant patients. They received two ml of normal saline intravenously as a placebo.

Group B: included 40 pregnant patients. They received (20mg) hyoscine butylbromide (one ml HBB+ one ml saline) intravenously.

Group C: included 40 pregnant patients .They received two ml (40 mg) hyoscine butylbromide intravenously (HBB).

DETAILED DESCRIPTION:
A case control trial Patients who meet the inclusion criteria were asked to participate in the study and a written consent was obtained from each patient after explaining thoroughly the nature and the scope of the study.

For each patient:

1. Complete history was taking to exclude allergy to hyoscine butylbromide, medical disorders with pregnancy (preeclampsia, diabetes mellitus, heart disease …etc.) and any contraindication for vaginal delivery.
2. General examination of the patients including (pulse, blood pressure, temperature).
3. Obstetric Abdominal examination including fetal lie, fetal presentation, head station and uterine contractions.
4. Vaginal examination including cervical dilatation, effacement and position, state of fetal membranes, presenting part, position of fetal head and pelvic adequacy.
5. Obstetric ultrasound to detect fetal gestational age, fetal birth weight amount of liquor, site of placental attachment and fetal heart rate.

Patients were divided into three equal groups:

Group A: included 40 pregnant patients. They received two ml of normal saline intravenously as a placebo.

Group B: included 40 pregnant patients. They received (20mg) hyoscine butylbromide (one ml HBB+ one ml saline) intravenously.

Group C: included 40 pregnant patients .They received two ml (40 mg) hyoscine butylbromide intravenously (HBB).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 35 years old
2. Primigravdae or multigravida
3. Gestational age between completed 37- 41 weeks + 6 days.
4. Uncomplicated cephalic singleton pregnancy occipto-anterior position.
5. Established spontaneous active labour (defined as the presence of at least three regular uterine contractions over 10 minutes with cervical dilatation three to four centimeters) with cervical effacement not less than 50%.
6. Intact amniotic membranes.
7. High risk pregnancy (women with pregnancy induced hypertension- cardiac-Diabetes Mellitus

Exclusion Criteria:

1. Multigravidae.
2. Multiple fetus.
3. Malpresentation.
4. Patients with indications of elective caesarean section.
5. Medical conditions associated with pregnancy e.g. preeclampsia, diabetes mellitus.
6. Contraindications for hyoscine butylbromide which include known allergy to hyoscine or other atropinics (e.g., atropine, scopolamine), myasthenia gravis, megacolon or glaucoma.
7. Patients presented to causality with spontaneous rupture of membranes.
8. Spontaneous rupture of membranes during the active phase of first stage of labour.
9. Oxytocin induction or augmentation.
10. Patients who underwent epidural anesthesia or other types of analgesia

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Actual)
Dates: Start 2017-02-11 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Duration of the first stage of labour | 24 hours
  Duration of the first stage of labour

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided